CLINICAL TRIAL: NCT00000347
Title: Risperidone for Treatment of Cocaine Dependence in Outpatients
Brief Title: Risperidone for Treatment of Cocaine Dependence in Outpatients - 12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-3-0010-12; Y01-3-0010-12
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1998-03

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this study is to evaluate pharmacological efficacy and clinical safety of risperidone in the treatment of cocaine and amphetamine dependence.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50 . Meet DSM-IV criteria for cocaine dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nuring women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical condtions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1997-07; Primary Completion 1998-08 (Actual); Study Completion 1998-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States